CLINICAL TRIAL: NCT06813924
Title: An Open-Label, Fixed-Sequence Study to Evaluate the Effect of Etavopivat on the Single-Dose Pharmacokinetics of Midazolam, Digoxin, Rosuvastatin, Pitavastatin, and Metformin in Healthy Adult Participants
Brief Title: A Research Study of the Effect of Etavopivat on Other Drugs in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7535-7976; U1111-1309-3456 (Other: Universal Trial Number)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers Sickle Cell Disease, Thalassemia
MeSH Terms: conditions — Thalassemia | interventions — Digoxin; pitavastatin; Metformin; Midazolam; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Period 1: digoxin+pitavastatin+metformin (Experimental): Participants will receive a single dose of oral digoxin, pitavastatin and metformin.
  Interventions: Drug: Digoxin; Drug: Pitavastatin; Drug: Metformin
- Period 1: midazolam+rosuvastatin (Experimental): Participants will receive a single dose of oral midazolam and rosuvastatin.
  Interventions: Drug: Midazolam; Drug: Rosuvastatin
- Period 2: etavopivat+midazolam (Experimental): Participants will receive a daily dose of oral etavopivat and single dose of oral midazolam.
  Interventions: Drug: Etavopivat; Drug: Midazolam
- Period 2: etavopivat+midazolam+rosuvastatin (Experimental): Participants will receive a daily dose of oral etavopivat, single dose of oral midazolam and rosuvastatin.
  Interventions: Drug: Etavopivat; Drug: Midazolam; Drug: Rosuvastatin
- Period 2: etavopivat+digoxin+pitavastatin+metformin (Experimental): Participants will receive a daily dose of oral etavopivat, single dose of oral digoxin, pitavastatin and metformin.
  Interventions: Drug: Etavopivat; Drug: Digoxin; Drug: Pitavastatin; Drug: Metformin

INTERVENTIONS:
Drug: Etavopivat — Participants will receive a daily dose of etavopivat orally.
  Arms: Period 2: etavopivat+digoxin+pitavastatin+metformin; Period 2: etavopivat+midazolam; Period 2: etavopivat+midazolam+rosuvastatin
Drug: Digoxin — Participants will receive a single dose of digoxin orally.
  Arms: Period 1: digoxin+pitavastatin+metformin; Period 2: etavopivat+digoxin+pitavastatin+metformin
Drug: Pitavastatin — Participants will receive a single dose of pitavastatin orally.
  Arms: Period 1: digoxin+pitavastatin+metformin; Period 2: etavopivat+digoxin+pitavastatin+metformin
Drug: Metformin — Participants will receive a single dose of metformin orally.
  Arms: Period 1: digoxin+pitavastatin+metformin; Period 2: etavopivat+digoxin+pitavastatin+metformin
Drug: Midazolam — Participants will receive a single dose of midazolam orally.
  Arms: Period 1: midazolam+rosuvastatin; Period 2: etavopivat+midazolam; Period 2: etavopivat+midazolam+rosuvastatin
Drug: Rosuvastatin — Participants will receive a single dose of rosuvastatin orally.
  Arms: Period 1: midazolam+rosuvastatin; Period 2: etavopivat+midazolam+rosuvastatin

SUMMARY:
The study aims to test if a new medicine called etavopivat potentially affects other medicines in healthy participants. The purpose of the study is to investigate whether the use of etavopivat affects the breakdown and metabolism of commonly used medicines in the body. During the study, participants will receive etavopivat and five different medicines that are already approved and available on the market, and which can be prescribed by doctors. These marketed medicines are called substrate drugs and they are: digoxin, pitavastatin, metformin, midazolam, and rosuvastatin. During a period of the study, participants will take 2 tablets of etavopivat daily for 10 consecutive days. The study will last for about 34 to 64 days.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 29.9 kilograms per square meter (kg/m^2) (both inclusive) at screening.
* Body weight greater than (>) 50.0 kg at screening.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to study interventions or related products.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive method.
* Exposure to an investigational medicinal product within 30 days or 5 half-lives of the investigational medicinal product (if known), whichever is longer, before screening.
* Participant is unable to refrain from or anticipates the use of any drug known to be a moderate or strong inhibitor or inducer of uridine 5'-diphospho-glucuronosyltransferase (UGT) enzymes, CYP3A4, CYP2C9, MATE1, OATP1B1/1B3, BCRP, OCT2, or P-gp, including St. John's Wort for 28 days prior to dosing and throughout the study.
* Use of any medication with unknown or unspecified content within 90 days before screening.
* Use of or intent to use prescription medicinal products or non-prescription drugs (including vitamins and herbal supplements) within 14 days prior to dosing and throughout the study, as declared by the participant, except for:
* Adequate contraceptive methods.
* Hormone replacement therapy (HRT) (for menopausal females).
* Over-the-counter topical medications known to not reach systemic circulation.
* Occasional use of acetaminophen up to 2 grams (g) (4 x 0.5 g) daily.
* Not able or not willing to adhere to study procedures, including:
* Eating the food provided in the study.
* Refraining from ingesting food or drinks that are not allowed during the study.
* Swallowing tablets.
* Abstaining from concomitant medication not allowed during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Cmax, digoxin, SD: Maximum observed digoxin plasma concentration with and without etavopivat at steady state | Day 1 and day 3 after digoxin administration
  Measured as picograms per milliliter (pg/mL).
AUC0-inf, digoxin, SD: Area under the digoxin plasma concentration-time curve from 0 hours and extrapolated to infinity with and without etavopivat at steady state | Day 1 and day 3 after digoxin administration
  Measured as hours*picograms per milliliter (h*pg/mL).
Cmax, rosuvastatin, SD: Maximum observed rosuvastatin plasma concentration with and without etavopivat at steady state | Day 1 after rosuvastatin administration
  Measured as pg/mL.
AUC0-inf, rosuvastatin, SD: Area under the rosuvastatin plasma concentration-time curve from 0 hours and extrapolated to infinity with and without etavopivat at steady state | Day 1 after rosuvastatin administration
  Measured as h*pg/mL.
Cmax, midazolam, SD: Maximum observed midazolam plasma concentration without etavopivat, with a single dose of etavopivat, and with etavopivat at steady state | Day 1 after midazolam administration
  Measured as pg/mL.
AUC0-inf, midazolam, SD: Area under the midazolam plasma concentration-time curve from 0 hours and extrapolated to infinity without etavopivat, with a single dose of etavopivat, and with etavopivat at steady state | Day 1 after midazolam administration
  Measured as h*pg/mL.
Cmax, pitavastatin, SD: Maximum observed pitavastatin plasma concentration with and without etavopivat at steady state | Day 1 and day 3 after pitavastatin administration
  Measured as nanograms per milliliter (ng/mL).
AUC0-inf, pitavastatin, SD: Area under the pitavastatin plasma concentration-time curve from 0 hours and extrapolated to infinity with and without etavopivat at steady state | Day 1 and day 3 after pitavastatin administration
  Measured as hours*nanograms per milliliter(h*ng/mL).
Cmax, metformin, SD: Maximum observed metformin plasma concentration with and without etavopivat at steady state | Day 1 and day 3 after metformin administration
  Measured as ng/mL.
AUC0-inf, metformin, SD: Area under the metformin plasma concentration-time curve from 0 hours and extrapolated to infinity with and without etavopivat at steady state | Day 1 and day 3 after metformin administration
  Measured as h*ng/mL.

SECONDARY OUTCOMES:
AUC0-last, digoxin, SD: Area under the digoxin plasma concentration-time curve from 0 hours to the last quantifiable concentration with and without etavopivat at steady state | Day 1 and day 3 after digoxin administration
  Measured as h*pg/mL.
t1/2, digoxin, SD: Terminal half-life for digoxin with and without etavopivat at steady state | Day 1 and day 3 after digoxin administration
  Measured as hours.
tmax, digoxin, SD: Time to maximum observed digoxin plasma concentration with and without etavopivat at steady state | Day 1 and day 3 after digoxin administration
  Measured as hours.
CL/Fdigoxin, SD: Apparent plasma clearance of digoxin with and without etavopivat at steady state | Day 1 and day 3 after digoxin administration
  Measured as liters per hour (L/h).
Vz/Fdigoxin, SD: Apparent volume of distribution of digoxin with and without etavopivat at steady state based on plasma concentration values | Day 1 and day 3 after digoxin administration
  Measured as liters (L).
AUC0-last, rosuvastatin, SD: Area under the rosuvastatin plasma concentration-time curve from 0 hours to the last quantifiable concentration with and without etavopivat at steady state | Day 1 after rosuvastatin administration
  Measured as h*pg/mL.
t1/2, rosuvastatin, SD: Terminal half-life for rosuvastatin with and without etavopivat at steady state | Day 1 after rosuvastatin administration
  Measured as hours.
tmax, rosuvastatin, SD: Time to maximum observed rosuvastatin plasma concentration with and without etavopivat at steady state | Day 1 after rosuvastatin administration
  Measured as hours.
CL/Frosuvastatin, SD: Apparent plasma clearance of rosuvastatin with and without etavopivat at steady state | Day 1 after rosuvastatin administration
  Measured as L/h.
Vz/Frosuvastatin, SD: Apparent volume of distribution of rosuvastatin with and without etavopivat at steady state based on plasma concentration values | Day 1 after rosuvastatin administration
  Measured as L.
AUC0-last, midazolam, SD: Area under the midazolam plasma concentration-time curve from 0 hours to the last quantifiable concentration without etavopivat, with a single dose of etavopivat, and with etavopivat at steady state | Day 1 after midazolam administration
  Measured as h*pg/mL.
t1/2, midazolam, SD: Terminal half-life for midazolam without etavopivat, with a single dose of etavopivat, and with etavopivat at steady state | Day 1 after midazolam administration
  Measured as hours.
tmax, midazolam, SD: Time to maximum observed midazolam plasma concentration without etavopivat, with a single dose of etavopivat, and with etavopivat at steady state | Day 1 after midazolam administration
  Measured as hours.
CL/Fmidazolam, SD: Apparent plasma clearance of midazolam without etavopivat, with a single dose of etavopivat and with etavopivat at steady state | Day 1 after midazolam administration
  Measured as L/h.
Vz/Fmidazolam, SD: Apparent volume of distribution of midazolam without etavopivat, with a single dose of etavopivat and with etavopivat at steady state | Day 1 after midazolam administration
  Measured as L.
AUC0-inf, 1-hydroxymidazolam, SD: Area under the midazolam plasma concentration-time curve from 0 hours and extrapolated to infinity without etavopivat, with a single dose of etavopivat, and with etavopivat at steady state | Day 1 after midazolam administration
  Measured as h*pg/mL.
Cmax, 1-hydroxymidazolam, SD: Maximum observed midazolam plasma concentration without etavopivat, with a single dose of etavopivat, and with etavopivat at steady state | Day 1 after midazolam administration
  Measured as pg/mL.
AUC0-last, 1-hydroxymidazolam, SD: Area under the midazolam plasma concentration-time curve from 0 hours to the last quantifiable concentration without etavopivat, with a single dose of etavopivat, and with etavopivat at steady state | Day 1 after midazolam administration
  Measured as h*pg/mL.
t1/2, 1-hydroxymidazolam: Terminal half-life for 1-hydroxymidazolam without etavopivat, with a single dose of etavopivat, and with etavopivat at steady state | Day 1 after midazolam administration
  Measured as hours.
tmax, 1-hydroxymidazolam: Time to maximum observed 1-hydroxymidazolam plasma concentration without etavopivat, with a single dose of etavopivat, and with etavopivat at steady state | Day 1 after midazolam administration
  Measured as hours.
CL/F1-hydroxymidazolam: Apparent plasma clearance of 1-hydroxymidazolam without etavopivat, with a single dose of etavopivat, and with etavopivat at steady state | Day 1 after midazolam administration
  Measured as L/h.
Vz/F1-hydroxymidazolam: Apparent volume of distribution of 1-hydroxymidazolam based on plasma concentration values without etavopivat, with a single dose of etavopivat, and with etavopivat at steady state | Day 1 after midazolam administration
  Measured as L.
AUC0-last, pitavastatin, SD: Area under the pitavastatin plasma concentration-time curve from 0 hours to the last quantifiable concentration with and without etavopivat at steady state | Day 1 and day 3 after pitavastatin administration
  Measured as h*ng/mL.
t1/2, pitavastatin, SD: Terminal half-life for pitavastatin with and without etavopivat at steady state | Day 1 and day 3 after pitavastatin administration
  Measured as hours.
tmax, pitavastatin, SD: Time to maximum observed pitavastatin plasma concentration with and without etavopivat at steady state | Day 1 and day 3 after pitavastatin administration
  Measured as hours.
CL/Fpitavastatin, SD: Apparent plasma clearance of pitavastatin with and without etavopivat at steady state | Day 1 and day 3 after pitavastatin administration
  Measured as L/h.
Vz/Fpitavastatin, SD: Apparent volume of distribution of pitavastatin with and without etavopivat at steady state based on plasma concentration values | Day 1 and day 3 after pitavastatin administration
  Measured as L.
AUC0-last, metformin, SD: Area under the metformin plasma concentration-time curve from 0 hours to the last quantifiable concentration with and without etavopivat at steady state | Day 1 and day 3 after metformin administration
  Measured as h*ng/mL.
t1/2, metformin, SD: Terminal half-life for metformin with and without etavopivat at steady state | Day 1 and day 3 after metformin administration
  Measured as hours.
tmax, metformin, SD: Time to maximum observed metformin plasma concentration with and without etavopivat at steady state | Day 1 and day 3 after metformin administration
  Measured as hours.
CL/Fmetformin, SD: Apparent plasma clearance of metformin with and without etavopivat at steady state | Day 1 and day 3 after metformin administration
  Measured as L/h.
Vz/Fmetformin, SD: Apparent volume of distribution of metformin with and without etavopivat at steady state based on plasma concentration values | Day 1 and day 3 after metformin administration
  Measured as L.
Aelast, metformin, SD%: Percentage of the metformin excreted into urine from the time of dosing to the collection time of the last measurable concentration with and without etavopivat at steady state | Day 1 and day 3 after metformin administration
  Measured as percentage (%) of the metformin excreted into urine.
CLR, metformin, SD: Renal clearance of metformin | Day 1 and day 3 after metformin administration
  Measured as L/h.
AUC0-tau, etavopivat: Area under the etavopivat plasma concentration-time curve during one dosing interval at single dose and at steady state | Day 1 and day 3 after etavopivat administration
  Measured as h*ng/mL.
AUC0-last etavopivat: Area under the etavopivat plasma concentration-time curve from 0 hours to the last quantifiable concentration at single dose and at steady state | Day 1 and day 3 after etavopivat administration
  Measured as h*ng/mL.
Cmax, etavopivat: Maximum observed etavopivat plasma concentration at single dose and at steady state | Day 1 and day 3 after etavopivat administration
  Measured as ng/mL.
t1/2, etavopivat: Terminal half-life for etavopivat at single dose and at steady state | Day 1 and day 3 after etavopivat administration
  Measured as hours.
tmax, etavopivat: Time to maximum observed etavopivat plasma concentration at single dose and at steady state | Day 1 and day 3 after etavopivat administration
  Measured as hours.
V/Fetavopivat: Apparent volume of distribution of etavopivat based on plasma concentration values at single dose and at steady state | Day 1 and day 3 after etavopivat administration
  Measured as L.
CL/Fetavopivat: Apparent plasma clearance of etavopivat at single dose and at steady state | Day 1 and day 3 after etavopivat administration
  Measured as L/h.
C, etavopivat: Observed etavopivat plasma concentration after single and multiple doses | From day 1 to day 4 after administration of etavopivat
  Measured as ng/mL.
Number of adverse events (AEs) | From first dose (day 1) until end of study (day 32)
  Measured as count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- ICON-Salt Lake City, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com